CLINICAL TRIAL: NCT03832452
Title: Prospective, Single-center, Randomized, Double-blind, Placebo-controlled, Two-part Phase 1 Study to Assess the Effect of Single Therapeutic and Supra-therapeutic Doses of Lucerastat on the QT/QTc Interval Duration in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Investigate Whether Administration of Lucerastat Can Affect Normal Heart Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-069-106; 2018-004546-42 (EudraCT Number)
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — migalastat; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized, double-blind, placebo-controlled, two-part Phase 1 study (Part A: parallel, 2 treatments; Part B: crossover, 4 treatments)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Treatment 1 (Experimental): A single oral dose of 2000 mg lucerastat on Day 1 and of 4000 mg lucerastat on Day 3
  Interventions: Drug: Lucerastat (Treatment A)
- Part A: Treatment 2 (Placebo Comparator): A single oral dose of placebo on Day 1 and 3
  Interventions: Other: Placebo
- Part B: Treatment A (Active Comparator): A single oral dose of 400 mg moxifloxacin
  Interventions: Drug: Moxifloxacin
- Part B: Treatment B (Experimental): A single oral dose of 1000 mg lucerastat
  Interventions: Drug: Lucerastat (Treatment B)
- Part B: Treatment C (Experimental): A single oral dose of 4000 mg lucerastat
  Interventions: Drug: Lucerastat (Treatment C)
- Part B: Treatment D (Placebo Comparator): A single oral dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lucerastat (Treatment A) — 2000 and 4000 mg; hard capsules for oral administration
  Arms: Part A: Treatment 1
Other: Placebo — hard capsules for oral administration
  Arms: Part A: Treatment 2; Part B: Treatment D
Drug: Moxifloxacin — 400 mg; film-coated tablets for oral administration
  Arms: Part B: Treatment A
Drug: Lucerastat (Treatment B) — 1000 mg; hard capsules for oral administration
  Arms: Part B: Treatment B
Drug: Lucerastat (Treatment C) — 4000 mg; hard capsules for oral administration
  Arms: Part B: Treatment C

SUMMARY:
Two-part Phase 1 study to assess the effect of single therapeutic and supra-therapeutic doses of lucerastat on the QT/QTc interval duration in healthy subjects (Part A: Pilot study; Part B: TQT study)

ELIGIBILITY:
Inclusion Criteria:

Part A only:

- Healthy male subjects aged between 18 and 55 years.

Part B only:

* Healthy male and female subjects aged between 18 and 55 years.
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 pre-dose of the first period. They must consistently and correctly use a highly effective method of contraception, or be sexually inactive, or have a vasectomized partner.
* Women of nonchildbearing potential (i.e., postmenopausal, XY genotype, Turner syndrome, uterine agenesis).

Part A and B:

* Signed informed consent prior to any study-mandated procedure.
* Body mass index of 18.0 to 30.0 kg/m2 (inclusive) at Screening. Body weight at least 50.0 kg at Screening and prior to first study treatment administration.
* Healthy on the basis of medical history, physical examination, cardiovascular assessments and clinical laboratory tests.

Exclusion Criteria:

Part B only:

* Known hypersensitivity to moxifloxacin or any of its excipients.
* Pregnant or lactating women.
* Women planning to become pregnant.

Part A and B:

* Previous exposure to lucerastat.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or presence of rhythm disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Part B: Placebo-corrected, change-from-baseline QTcF (ΔΔQTcF) | From 1 h pre-dose to 36 hour after study treatment administration (duration: up to 37 hours)
  QTcF = QT interval corrected with Fridericia's formula; ΔΔQTcF = Placebo-corrected change-from-baseline QTcF

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller MS, Sidharta PN, Voors-Pette C, Darpo B, Xue H, Dingemanse J. The effect of the glucosylceramide synthase inhibitor lucerastat on cardiac repolarization: results from a thorough QT study in healthy subjects. Orphanet J Rare Dis. 2020 Oct 27;15(1):303. doi: 10.1186/s13023-020-01582-7. PMID 33109218